CLINICAL TRIAL: NCT02155868
Title: Cerebral Near-Infrared Spectroscopy Monitoring in High-Risk Cardiac Surgery Patients: A Prospective, Randomised, Single-Blinded Study
Brief Title: Role of Cerebral Oximetry in Reducing Postoperative Morbidity Following Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Evgeny Fominskiy, MD, PhD, Mr, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIRS-in-CS
Record Dates: First submitted 2014-05-31; First posted 2014-06-04 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Complications
Keywords: Cerebral near-infrared spectroscopy monitoring; Postoperative complications; Cardiac surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Cerebral NIRS monitoring by means of FORE-SIGHT Universal Cerebral Oximeter MC-2030C.
  Predefined protocol of interventions for correcting rSO2 desaturation (< 60%) during cardiac surgery and the first six hours after it.
  Interventions: Other: Correction rSO2 desaturation.
- Control (Placebo Comparator): Only cerebral NIRS monitoring by means of FORE-SIGHT Universal Cerebral Oximeter MC-2030C during cardiac surgery and the first six hours after it.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Correction rSO2 desaturation. — Predefined protocol of interventions for correcting rSO2 desaturation (< 60%) during cardiac surgery and the first six hours after it.
  In case of rSO2 decrease less than 60% correct:
  head position; position of aortic,venous cannulae and central venous catheters; partial pressure of carbon dioxide in arterial blood < 35 mmHg; mean arterial pressure < 60 mmHg; central venous pressure > 10 mmHg; cardiac index < 2.0 l/min/m2; mixed venous oxygen saturation < 60%; hemoglobin < 65 g/L during cardiopulmonary bypass or hemoglobin < 90 g/L after cardiopulmonary bypass; decrease cerebral O2 consumption.
  Arms: Intervention
Other: Standard treatment — Standard treatment
  Arms: Control

SUMMARY:
Cerebral oximetry employing near-infrared spectroscopy (NIRS) is a non-invasive modality used to estimate regional cerebral oxygen content saturation (rSO2). Near-infrared spectroscopy has increasingly been used in perioperative setting of heart surgery and many studies have outlined an increased incidence of postoperative morbidity in patients with significant perioperative reductions in rSO2. Although a relationship between rSO2 reductions and adverse outcomes has been reported, there is not compelling evidence that interventions to correct rSO2 during cardiac surgery lead to improved clinical outcomes.

Hypothesis of the study is that interventions to normalize intraoperatively decreased cerebral rSO2 would reduce the overall incidence of postoperative complications in high-risk cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

High-risk cardiac surgery patients as determined by at least one of the followings:

* the age greater than or equal to 75 years on the day of screening;
* left ventricle ejection fraction less than 35%;
* use of a preoperative intraaortic balloon pump;
* combined valve and coronary artery surgery or multiple valve surgery in patients who have congestive heart failure, or renal insufficiency (creatinine clearance < 60 ml/min)

Exclusion Criteria:

* refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative complications | Up to 30 day after randomisation
  This composite outcome includes: myocardial infarction, stroke, delirium, postoperative cognitive dysfunction, wound infection, mediastinitis, mechanical ventilation more than 24 h, arrhythmia, reoperation for bleeding, acute kidney injury, and acute kidney injury requiring dialysis.

SECONDARY OUTCOMES:
Incidence of major organ morbidity and mortality | Up to 30 day after randomization
  This outcome includes: stroke, acute kidney injury requiring dialysis, mechanical ventilation more than 48 h, mediastinitis, reoperation, and death
Duration of intensive care unit stay | Up to 30 day after randomization
Duration of postoperative hospital stay | Up to 30 day after randomization
Death from all causes at 30 days | Up to 30 day after randomisation

OTHER OUTCOMES:
Incidence of desaturation episodes | Intra operative
  Desaturation is defined as level of rSO2 less than 60%.
Severity of desaturation episodes | Intra operative
  Severity is defined as the product of length of time and depth of rSO2 less than 60%

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Lomivorotov, Prof, Principal Investigator — Academician EN Meshalkin Novosibirsk State Budget Research Institute of Circulation Pathology
Locations (1):
- Academician EN Meshalkin Novosibirsk State Budget Research Institute of Circulation Pathology, Novosibirsk, Novosibirsk Territory, Russia

REFERENCES:
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Yao FS, Tseng CC, Ho CY, Levin SK, Illner P. Cerebral oxygen desaturation is associated with early postoperative neuropsychological dysfunction in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Oct;18(5):552-8. doi: 10.1053/j.jvca.2004.07.007. PMID 15578464
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Background] Fischer GW, Lin HM, Krol M, Galati MF, Di Luozzo G, Griepp RB, Reich DL. Noninvasive cerebral oxygenation may predict outcome in patients undergoing aortic arch surgery. J Thorac Cardiovasc Surg. 2011 Mar;141(3):815-21. doi: 10.1016/j.jtcvs.2010.05.017. Epub 2010 Jun 25. PMID 20579669
- [Background] Heringlake M, Garbers C, Kabler JH, Anderson I, Heinze H, Schon J, Berger KU, Dibbelt L, Sievers HH, Hanke T. Preoperative cerebral oxygen saturation and clinical outcomes in cardiac surgery. Anesthesiology. 2011 Jan;114(1):58-69. doi: 10.1097/ALN.0b013e3181fef34e. PMID 21178669
- [Background] Denault A, Deschamps A, Murkin JM. A proposed algorithm for the intraoperative use of cerebral near-infrared spectroscopy. Semin Cardiothorac Vasc Anesth. 2007 Dec;11(4):274-81. doi: 10.1177/1089253207311685. PMID 18270192